CLINICAL TRIAL: NCT01408589
Title: A Pharmacotherapy Study: A Dose Response Effect of Atomoxetine on Alcohol-elicited Craving and Sensitivity to the Acute Effects of Alcohol
Brief Title: A Dose Response Effect of Atomoxetine to the Acute Effects of Alcohol
Acronym: ATX_COMT
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: University of Colorado, Boulder (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH); National Center for Research Resources (NCRR) (NIH)
Responsible Party: Heather M. Haughey, P.I., University of Colorado, Boulder
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: B5089; K01AA015331 (NIH); M01RR000051 (NIH)
Record Dates: First submitted 2011-07-12; First posted 2011-08-03 (Estimated); Last update posted 2011-08-03 (Estimated); Status verified 2011-08

CONDITIONS: Alcohol Craving; Mood Changes
Keywords: alcohol; craving; mood; optimum dose of atomoxetine
MeSH Terms: interventions — Atomoxetine Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Sugar Pill (Placebo Comparator)
  Interventions: Drug: Atomoxetine, Strattera
- Atomoxetine 40 mg (Experimental)
  Interventions: Drug: Atomoxetine, Strattera
- Atomoxetine 60 mg (Experimental)
  Interventions: Drug: Atomoxetine, Strattera
- Atomoxetine 80 mg (Experimental)
  Interventions: Drug: Atomoxetine, Strattera

INTERVENTIONS:
Drug: Atomoxetine, Strattera — Atomoxetine at 0, 40, 60, 80 mg/day was given for 5 days, all subjects took two capsules per day for 5 days; all active dose groups received 40 mg/day for first 3 days and where then dose escalated to dosage group assigned.

SUMMARY:
This two-stage study will examine the effects of a 5 day course of atomoxetine (placebo, 40, 60 or 80 mg/day; Strattera) (a selective NE transporter (NET) inhibitor) on alcohol-elicited craving and sensitivity to alcohol. The novelty of this study is that of atomoxetine and the fact that it targets NET, neither of which has heretofore been examined in the context of alcohol dependence. It is hopeful that this pilot study, of 86 total individuals, will provide the PI with sufficient preliminary data to submit a subsequent R01 application to study atomoxetine and the involvement of specific single nucleotide polymorphisms within the NET gene on alcohol-related phenotypes in alcohol dependent and non-dependent populations. The long-term objective of this research is to develop more efficacious treatment interventions for alcohol abuse and dependence.

Hypothesis 1: It is hypothesized that subjects who receive 40, 60 or 80 mg/day of atomoxetine for 5 days will demonstrate significantly less alcohol-elicited craving than subjects who receive a placebo.

Hypothesis 2: It is hypothesized that subjects who receive 40, 60 or 80 mg/day of atomoxetine for 5 days will be less sensitive to the acute effects of alcohol (subjective intoxication) than subjects who receive a placebo.

ELIGIBILITY:
Inclusion Criterion:

1. Males and females age 21 to 35, as verified upon the presentation of a valid driver's license;
2. Must drink alcohol at least twice a week and have a minimum of 3 drinks per occasion (2 for women);
3. Must score 8 or higher on the Alcohol Use Disorders Identification Test (AUDIT; Babor et al., 1992). The AUDIT is a screening instrument used to identify persons whose alcohol consumption is characterized by moderate to heavy drinking;
4. No history of alcohol treatment or desire for treatment;
5. Not currently take medications that are contraindicated for concurrent use with alcohol;
6. Female subjects must not be pregnant, as indicated by a pregnancy test that will be conducted immediately prior dispensing of medication.

Exclusion Criterion:

Subjects who have hypertension, tachycardia, cardiovascular disease, hepatic or renal impairment, pregnant or who are currently using MAO inhibitors, Albuterol or other pressor agents will be excluded from this study.

Ages: 21 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 86 (Actual)
Dates: Start 2005-06; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Alcohol Craving | Day 5 of medication
  Alcohol craving and sensitivity were measured with the AUQ, ARS, POMS, BAES and SHAS

SECONDARY OUTCOMES:
Genetic moderation | day 5 of medication
  To determine whether two functional SNPs within the COMT and DBH genes moderate the effects of EtOH and or atomoxetine.
  COMT Val158Met (G/A), Val > Met 2-4x plasma activity DBH -1021 C/T, C/C has 3x more plasma activity NET gene variants were also examined

CONTACTS AND LOCATIONS:
Overall Officials: Heather M Haughey, Ph.D., Principal Investigator — University of Colorado, Boulder
Locations (1):
- GCRC, University of Colorado Boulder, Boulder, Colorado, United States